CLINICAL TRIAL: NCT00648960
Title: Single Dose Crossover Comparative Bioavailability Study of Clarithromycin 500 mg Tablets in Healthy Male and Female Volunteers / Fasting State
Brief Title: Comparative Bioavailability Study of Clarithromycin 500 mg Tablets in Fasting State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Collaborators: Genpharm ULC (Industry)
Responsible Party: Elliot Offman Director, Biopharmaceutics, Genpharm ULC
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAI-P3-134
Record Dates: First submitted 2008-03-31; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Clarithromycin
- 2 (Active Comparator)
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Single-dose 500 mg immediate-release oral tablet
  Arms: 1
Drug: Clarithromycin — Single-dose 500 mg immediate-release oral dose
  Other Names: Biaxin®; Biaxin® Filmtabs
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Genpharm's clarithromycin tablets following a single, oral 500 mg (1 x 500 mg) dose compared to the Biaxin® filmtab® (Abbott Laboratories USA) administered under fasting conditions. Sixty-four (64) healthy, light-, non- or ex-smoking subjects of at least 18 a years of age were randomized, in this two-period, two-treatment crossover bioequivalence study conducted by Eric Sicard, M.D. at Algorithme Pharma Inc. Montreal, Canada.

Statistical analysis of the data reveals that 90% confidence intervals are within the acceptable bioequivalent range of 80% and 125% for the natural log transformed parameters AUCT, AUCI and Cmax. This study demonstrates that Genpharm's clarithromycin 500 mg tablets are bioequivalent to Biaxin® filmtab® 500 mg tablets (Abbott Laboratories USA) administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria may be included in the study:

Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form duly signed by the subject

Males or females aged from 18 to 55 years with a body mass index (BMI) greater than or equal to 19 and below 30; demographic data (sex, age, ethnic group, body weight, height and smoking habits) will be recorded and reported in the final report

Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance and must be recorded as such in the CRF (laboratory tests are presented in section 7.1.3)

Healthy according to the laboratory results and physical examination

Exclusion Criteria:

Significant history of hypersensitivity to clarithromycin, erythromycin, other macrolide antibacterial agents or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs

Presence or history of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects

Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease

Females who are pregnant, lactating or are likely to become pregnant during the study phases

Females of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the study

Positive pregnancy test before or during the study

Use of the following products (astemizole, terfenadine, cisapride or pimozide) in the previous 14 days before day 1 of the study

Maintenance therapy with any drug, or significant history of drug dependency, alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic), or serious psychological disease

Any clinically significant illness in the previous 28 days before day 1 of this study

Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.)

Participation in another clinical trial in the previous 28 days before day 1 of this study

Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Positive urine screening of drugs of abuse (drug names are presented in section 7.1.4)

Positive results to HIV, HBsAg or anti-HCV tests

History of fainting upon blood sampling

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2003-07; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic; The 90% confidence interval for the exponential of the difference between the Test and the Reference product for the ln-transformed parameters Cmax, AUCT and AUC∞ should be between 80 and 125%. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Laval, Quebec, Canada

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html